CLINICAL TRIAL: NCT05677113
Title: A Phase II Study of Perioperative QBECO Site Specific Immunomodulator (Qu Biologics®) in Patients With Metastatic Colorectal Adenocarcinoma Within the Liver Undergoing Resection
Brief Title: A Study of QBECO Versus Placebo in the Treatment of Colorectal Cancer That Has Spread to the Liver
Acronym: PERIOP-06
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 4023
Record Dates: First submitted 2022-11-04; First posted 2023-01-10 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2024-03

CONDITIONS: Colorectal Cancer; Liver Metastases
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- QBECO (Experimental): QBECO is an SSI formulated from inactivated E. coli bacteria that is specifically designed to target pathologies of the gastrointestinal (GI) tract and related organs, such as the liver. This trial will test the hypothesis that in patients undergoing resection of colorectal liver metastases (CRLMs), perioperative treatment with QBECO will attenuate the postoperative immune suppression and will improve progression-free survival (PFS).
  Interventions: Drug: QBECO
- Placebo (Placebo Comparator): A placebo is a liquid that looks like the study drug, but contains no medication.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: QBECO — QBECO is a site specific immunomodulator (SSI) designed to promote innate immune responses in the gastrointestinal tract and related organs, including the liver. QBECO will be administered according to the following regimen: 0.1mL self-administered subcutaneous injections every 2 days for 11-120 days preoperatively, and 41 days postoperatively.
  Arms: QBECO
Drug: Placebo — Placebo will be prepared in the same way as the IP. Placebo will be administered according to the following regimen: 0.1mL self-administered subcutaneous injections every 2 days for 11-120 days preoperatively, and 41 days postoperatively.
  Arms: Placebo

SUMMARY:
The goal of this type of clinical trial is t to answer the following question: Can the chance of colorectal cancer progressing be lowered by taking a medication, QBECO, before and after surgery? The goal of this study is to find out if this approach is better or worse than the standard of care for your type of cancer. The standard of care is defined as care most people get for metastatic colorectal cancer. There is currently no standard of care drug being given before or after surgery to prevent further spread of your cancer. Participants will be asked to self-inject the study medication before surgery for minimum of 11 days and after surgery for minimum of 41 days. Participants will be followed up every 3 months for 2 years, with a final visit at year 5.

DETAILED DESCRIPTION:
PERIOP-06 is a multicenter, phase II, blinded, randomized, placebo-controlled trial in adult patients planned to undergo resection of colorectal liver metastases (CRLM) for complete clearance of all visible disease. The investigational product for the study is QBECO. QBECO is a site specific immunomodulator (SSI) designed to promote innate immune responses in the gastrointestinal tract and related organs, including the liver. This trial is motivated by the promising preclinical and clinical data supporting the safety and efficacy of QBECO in attenuating postoperative immunosuppression and the resulting proliferation of cancer.

The primary objective of this randomized controlled trial is to determine if QBECO administered perioperatively can improve 2-year Progression-Free Survival in adult patients undergoing resection of CRLMs for complete clearance of metastatic disease. The main secondary objectives will be to:

1. Determine the effect of QBECO on the frequency and kinetics of clearance (and recurrence) of circulating tumor DNA (ctDNA) in the postoperative period and further evaluate the use ctDNA as part of ongoing surveillance.
2. Determine the side-effect profile of perioperative QBECO.
3. Determine the effect of QBECO on 5-year overall survival

Approximately 115 participants will be randomized to receive a placebo or the investigational product, QBECO. QBECO or placebo will be administered according to the following regimen: 0.1mL subcutaneous injections every two days for 11-120 days preoperatively, and 41 days postoperatively. Participants will be followed for 5 years after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older at time of enrollment.
* Pathologic diagnosis of colorectal carcinoma with clinical diagnosis of liver metastases
* Planned to undergo resection of liver lesions for complete clearance of all visible metastatic disease. This will include those who may undergo synchronous resection of the primary colorectal cancer and/or those who may receive a combination of surgery and ablation to treat all lesions.
* Computerized Tomography (CT) of the chest, abdomen, and pelvis with intravenous (IV) contrast within 6 weeks prior to enrollment.
* MRI of the liver within 6 weeks prior to enrollment OR within 6 weeks prior to starting neoadjuvant chemotherapy (for patients treated with chemotherapy).
* Planned to receive the last dose of neoadjuvant chemotherapy at least 25 days prior to surgery (for patients treated with neoadjuvant chemotherapy).
* Agree to comply with the contraceptive requirements of the protocol when applicable
* Willing and able to either perform subcutaneous injections according to the study protocol, or receive the injections from a caregiver delegated by the participant.
* Able to provide informed consent or has a substitute decision maker capable of providing consent on their behalf.

Exclusion Criteria:

* Prior or current evidence of extrahepatic metastases. Patients with small (<1.0 cm) indeterminate pulmonary nodules may be included at the investigator's discretion.
* Prior hepatic arterial infusion or embolization. Prior portal vein embolization, ablation, or liver resection are permitted.
* Patients with any invasive cancer history other than colorectal cancer in the last 5 years. In situ disease (e.g., melanoma in situ, ductal carcinoma in situ of the breast) or non melanoma skin cancers are permitted.
* Patients with a documented history of clinically severe autoimmune disease or a syndrome that requires systemic steroids or immunosuppressive agents. This includes patient requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent, or depot corticosteroids in the 6 weeks before enrollment) or immunosuppressant drugs (such as azathioprine, tacrolimus, cyclosporine, etc.) within the 14 days prior to enrollment or a reasonable expectation that the patient may require such treatment during the course of the study. Inhaled or topical or inter-articular steroids, and adrenal replacement steroid doses ≤ 10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease. Steroids used for premedication prior to chemotherapy or as part of a chemotherapy regimen are allowed.
* Patients with known active human immunodeficiency virus (HIV), Hepatitis B, or Hepatitis C infections.
* Pregnant patients or those who are nursing an infant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Estimated)
Dates: Start 2023-08-30 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2030-02-01 (Estimated)

PRIMARY OUTCOMES:
The primary outcome will be the 2-year Progression-Free Survival (PFS) rate | 2 years
  PFS will be defined as the time from enrollment to the first event that is either locoregional recurrence (of the resected primary colorectal adenocarcinoma or the resected ± intraoperatively ablated metastatic disease), distant metastases, or death from any cause.
  Section 5 further defines PFS and its measurement.

SECONDARY OUTCOMES:
Clearance of ctDNA. | 5 years
  A substantial body of research has demonstrated associations between ctDNA and cancer progression.Timing of measurement will be at baseline (which will occur within 14 days prior to the first dose of Investigational Product (IP) and at least 14 days after the last dose of chemotherapy, when applicable), preoperatively on the day of surgery, and postoperatively. A sample of fresh tumour tissue will be obtained from each resected hepatic and extrahepatic (when applicable) tumour site, resection of the primary colorectal carcinoma, along with a sample of normal adjacent tissue (one per surgical specimen) to tailor the ctDNA assay to the individual participant's tumour profile. If tumour tissue is not available from the resected specimen, tumour tissue from a prior resection or biopsy of the participant's adenocarcinoma may be requested. If disease progression is detected, ctDNA will also be measured at that time.
Side-effect profile of QBECO | through study completion, an average of 5 years
  This will include an evaluation of AEs and postoperative complications in the treatment and control groups. A postoperative complication will be defined as any deviation from the normal postoperative course. All clearly related signs, symptoms, and abnormal diagnostic procedures should be recorded in the source document and should be grouped under one diagnosis. The deviation must be possibly or probably related to the surgery and must occur postoperatively. The modified Clavien-Dindo system will be used to define and classify postoperative complications.
Quality of recovery | Baseline; postoperative day 3, and 6 weeks postoperatively
  Measured by the QoR-40. The QoR-40 is a validated tool designed to measure the early postoperative health status of patients. The tool has been widely used as a patient-reported outcome measure of recovery after surgery and has been translated into multiple languages. Timing of measurement will be at baseline (which will occur within 14 days prior to the first IP dose and at least 14 days after the last dose of chemotherapy, when applicable), on postoperative day (POD) 3, and 6 weeks postoperatively. The survey may be administered in person or virtually by telephone or video call.
Five-year overall survival | 5 years
  This will be measured from date of enrollment to the date of death.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Karanicolas, Principal Investigator — Paul.Karanicolas@sunnybrook.ca
Locations (4):
- Canada (4):
  - Hamilton Health Science Centre, Hamilton, Ontario
  - London Health Science Centre, London, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Sunnybrook Health Science Centre, Toronto, Ontario

REFERENCES:
- [Background] Tsuchiya Y, Sawada S, Yoshioka I, Ohashi Y, Matsuo M, Harimaya Y, Tsukada K, Saiki I. Increased surgical stress promotes tumor metastasis. Surgery. 2003 May;133(5):547-55. doi: 10.1067/msy.2003.141. PMID 12773983
- [Background] Tai LH, Zhang J, Scott KJ, de Souza CT, Alkayyal AA, Ananth AA, Sahi S, Adair RA, Mahmoud AB, Sad S, Bell JC, Makrigiannis AP, Melcher AA, Auer RC. Perioperative influenza vaccination reduces postoperative metastatic disease by reversing surgery-induced dysfunction in natural killer cells. Clin Cancer Res. 2013 Sep 15;19(18):5104-15. doi: 10.1158/1078-0432.CCR-13-0246. Epub 2013 Jul 23. PMID 23881927
- [Background] Tai LH, Alkayyal AA, Leslie AL, Sahi S, Bennett S, Tanese de Souza C, Baxter K, Angka L, Xu R, Kennedy MA, Auer RC. Phosphodiesterase-5 inhibition reduces postoperative metastatic disease by targeting surgery-induced myeloid derived suppressor cell-dependent inhibition of Natural Killer cell cytotoxicity. Oncoimmunology. 2018 Mar 1;7(6):e1431082. doi: 10.1080/2162402X.2018.1431082. eCollection 2018. PMID 29872554
- [Background] Tai LH, de Souza CT, Belanger S, Ly L, Alkayyal AA, Zhang J, Rintoul JL, Ananth AA, Lam T, Breitbach CJ, Falls TJ, Kirn DH, Bell JC, Makrigiannis AP, Auer RA. Preventing postoperative metastatic disease by inhibiting surgery-induced dysfunction in natural killer cells. Cancer Res. 2013 Jan 1;73(1):97-107. doi: 10.1158/0008-5472.CAN-12-1993. Epub 2012 Oct 22. PMID 23090117
- [Background] Seth R, Tai LH, Falls T, de Souza CT, Bell JC, Carrier M, Atkins H, Boushey R, Auer RA. Surgical stress promotes the development of cancer metastases by a coagulation-dependent mechanism involving natural killer cells in a murine model. Ann Surg. 2013 Jul;258(1):158-68. doi: 10.1097/SLA.0b013e31826fcbdb. PMID 23108132
- [Background] Ananth AA, Tai LH, Lansdell C, Alkayyal AA, Baxter KE, Angka L, Zhang J, Tanese de Souza C, Stephenson KB, Parato K, Bramson JL, Bell JC, Lichty BD, Auer RC. Surgical Stress Abrogates Pre-Existing Protective T Cell Mediated Anti-Tumor Immunity Leading to Postoperative Cancer Recurrence. PLoS One. 2016 May 19;11(5):e0155947. doi: 10.1371/journal.pone.0155947. eCollection 2016. PMID 27196057
- [Background] Gabrilovich DI. Myeloid-Derived Suppressor Cells. Cancer Immunol Res. 2017 Jan;5(1):3-8. doi: 10.1158/2326-6066.CIR-16-0297. PMID 28052991
- [Background] Manz MG, Boettcher S. Emergency granulopoiesis. Nat Rev Immunol. 2014 May;14(5):302-14. doi: 10.1038/nri3660. Epub 2014 Apr 22. PMID 24751955
- [Background] Angka L, Martel AB, Kilgour M, Jeong A, Sadiq M, de Souza CT, Baker L, Kennedy MA, Kekre N, Auer RC. Natural Killer Cell IFNgamma Secretion is Profoundly Suppressed Following Colorectal Cancer Surgery. Ann Surg Oncol. 2018 Nov;25(12):3747-3754. doi: 10.1245/s10434-018-6691-3. Epub 2018 Sep 5. PMID 30187278
- [Background] Zhang J, Tai LH, Ilkow CS, Alkayyal AA, Ananth AA, de Souza CT, Wang J, Sahi S, Ly L, Lefebvre C, Falls TJ, Stephenson KB, Mahmoud AB, Makrigiannis AP, Lichty BD, Bell JC, Stojdl DF, Auer RC. Maraba MG1 virus enhances natural killer cell function via conventional dendritic cells to reduce postoperative metastatic disease. Mol Ther. 2014 Jul;22(7):1320-1332. doi: 10.1038/mt.2014.60. Epub 2014 Apr 3. PMID 24695102
- [Background] Mitroulis I, Ruppova K, Wang B, Chen LS, Grzybek M, Grinenko T, Eugster A, Troullinaki M, Palladini A, Kourtzelis I, Chatzigeorgiou A, Schlitzer A, Beyer M, Joosten LAB, Isermann B, Lesche M, Petzold A, Simons K, Henry I, Dahl A, Schultze JL, Wielockx B, Zamboni N, Mirtschink P, Coskun U, Hajishengallis G, Netea MG, Chavakis T. Modulation of Myelopoiesis Progenitors Is an Integral Component of Trained Immunity. Cell. 2018 Jan 11;172(1-2):147-161.e12. doi: 10.1016/j.cell.2017.11.034. PMID 29328910
- [Background] Kaufmann E, Sanz J, Dunn JL, Khan N, Mendonca LE, Pacis A, Tzelepis F, Pernet E, Dumaine A, Grenier JC, Mailhot-Leonard F, Ahmed E, Belle J, Besla R, Mazer B, King IL, Nijnik A, Robbins CS, Barreiro LB, Divangahi M. BCG Educates Hematopoietic Stem Cells to Generate Protective Innate Immunity against Tuberculosis. Cell. 2018 Jan 11;172(1-2):176-190.e19. doi: 10.1016/j.cell.2017.12.031. PMID 29328912
- [Background] Netea MG, Joosten LAB, van der Meer JWM. Hypothesis: stimulation of trained immunity as adjunctive immunotherapy in cancer. J Leukoc Biol. 2017 Dec;102(6):1323-1332. doi: 10.1189/jlb.5RI0217-064RR. Epub 2017 Oct 10. PMID 29018149
- [Background] Bazett M, Costa AM, Bosiljcic M, Anderson RM, Alexander MP, Wong SWY, Dhanji S, Chen JM, Pankovich J, Lam S, Sutcliffe S, Gunn H, Kalyan S, Mullins DW. Harnessing innate lung anti-cancer effector functions with a novel bacterial-derived immunotherapy. Oncoimmunology. 2017 Nov 27;7(3):e1398875. doi: 10.1080/2162402X.2017.1398875. eCollection 2018. PMID 29399400
- [Background] Kalyan S, Bazett M, Sham HP, Bosiljcic M, Luk B, Dhanji S, Costa AM, Wong SWY, Netea MG, Mullins DW, Gunn H. Distinct inactivated bacterial-based immune modulators vary in their therapeutic efficacies for treating disease based on the organ site of pathology. Sci Rep. 2020 Apr 3;10(1):5901. doi: 10.1038/s41598-020-62735-z. PMID 32246043
- [Background] Faraj TA, McLaughlin CL, Erridge C. Host defenses against metabolic endotoxaemia and their impact on lipopolysaccharide detection. Int Rev Immunol. 2017 May 4;36(3):125-144. doi: 10.1080/08830185.2017.1280483. Epub 2017 Mar 1. PMID 28783409
- [Background] Sham HP, Bazett M, Bosiljcic M, Yang H, Luk B, Law HT, Morampudi V, Yu HB, Pankovich J, Sutcliffe S, Bressler B, Marshall JK, Fedorak RN, Chen J, Jones M, Gunn H, Kalyan S, Vallance BA. Immune Stimulation Using a Gut Microbe-Based Immunotherapy Reduces Disease Pathology and Improves Barrier Function in Ulcerative Colitis. Front Immunol. 2018 Sep 27;9:2211. doi: 10.3389/fimmu.2018.02211. eCollection 2018. PMID 30319652
- [Background] Sutcliffe S, Kalyan S, Pankovich J, Chen JMH, Gluck R, Thompson D, Bosiljcic M, Bazett M, Fedorak RN, Panaccione R, Axler J, Marshall JK, Mullins DW, Kabakchiev B, McGovern DPB, Jang J, Coldman A, Vandermeirsch G, Bressler B, Gunn H. Novel Microbial-Based Immunotherapy Approach for Crohn's Disease. Front Med (Lausanne). 2019 Jul 19;6:170. doi: 10.3389/fmed.2019.00170. eCollection 2019. PMID 31380382
- [Background] Hackl C, Neumann P, Gerken M, Loss M, Klinkhammer-Schalke M, Schlitt HJ. Treatment of colorectal liver metastases in Germany: a ten-year population-based analysis of 5772 cases of primary colorectal adenocarcinoma. BMC Cancer. 2014 Nov 4;14:810. doi: 10.1186/1471-2407-14-810. PMID 25369977
- [Background] Manfredi S, Lepage C, Hatem C, Coatmeur O, Faivre J, Bouvier AM. Epidemiology and management of liver metastases from colorectal cancer. Ann Surg. 2006 Aug;244(2):254-9. doi: 10.1097/01.sla.0000217629.94941.cf. PMID 16858188
- [Background] Engstrand J, Nilsson H, Stromberg C, Jonas E, Freedman J. Colorectal cancer liver metastases - a population-based study on incidence, management and survival. BMC Cancer. 2018 Jan 15;18(1):78. doi: 10.1186/s12885-017-3925-x. PMID 29334918
- [Background] Nordlinger B, Sorbye H, Glimelius B, Poston GJ, Schlag PM, Rougier P, Bechstein WO, Primrose JN, Walpole ET, Finch-Jones M, Jaeck D, Mirza D, Parks RW, Collette L, Praet M, Bethe U, Van Cutsem E, Scheithauer W, Gruenberger T; EORTC Gastro-Intestinal Tract Cancer Group; Cancer Research UK; Arbeitsgruppe Lebermetastasen und-tumoren in der Chirurgischen Arbeitsgemeinschaft Onkologie (ALM-CAO); Australasian Gastro-Intestinal Trials Group (AGITG); Federation Francophone de Cancerologie Digestive (FFCD). Perioperative chemotherapy with FOLFOX4 and surgery versus surgery alone for resectable liver metastases from colorectal cancer (EORTC Intergroup trial 40983): a randomised controlled trial. Lancet. 2008 Mar 22;371(9617):1007-16. doi: 10.1016/S0140-6736(08)60455-9. PMID 18358928
- [Background] Portier G, Elias D, Bouche O, Rougier P, Bosset JF, Saric J, Belghiti J, Piedbois P, Guimbaud R, Nordlinger B, Bugat R, Lazorthes F, Bedenne L. Multicenter randomized trial of adjuvant fluorouracil and folinic acid compared with surgery alone after resection of colorectal liver metastases: FFCD ACHBTH AURC 9002 trial. J Clin Oncol. 2006 Nov 1;24(31):4976-82. doi: 10.1200/JCO.2006.06.8353. PMID 17075115
- [Background] Kanemitsu Y, Shimizu Y, Mizusawa J, Inaba Y, Hamaguchi T, Shida D, Ohue M, Komori K, Shiomi A, Shiozawa M, Watanabe J, Suto T, Kinugasa Y, Takii Y, Bando H, Kobatake T, Inomata M, Shimada Y, Katayama H, Fukuda H; JCOG Colorectal Cancer Study Group. Hepatectomy Followed by mFOLFOX6 Versus Hepatectomy Alone for Liver-Only Metastatic Colorectal Cancer (JCOG0603): A Phase II or III Randomized Controlled Trial. J Clin Oncol. 2021 Dec 1;39(34):3789-3799. doi: 10.1200/JCO.21.01032. Epub 2021 Sep 14. PMID 34520230
- [Background] Oxnard GR, Paweletz CP, Kuang Y, Mach SL, O'Connell A, Messineo MM, Luke JJ, Butaney M, Kirschmeier P, Jackman DM, Janne PA. Noninvasive detection of response and resistance in EGFR-mutant lung cancer using quantitative next-generation genotyping of cell-free plasma DNA. Clin Cancer Res. 2014 Mar 15;20(6):1698-1705. doi: 10.1158/1078-0432.CCR-13-2482. Epub 2014 Jan 15. PMID 24429876
- [Background] Goldberg SB, Narayan A, Kole AJ, Decker RH, Teysir J, Carriero NJ, Lee A, Nemati R, Nath SK, Mane SM, Deng Y, Sukumar N, Zelterman D, Boffa DJ, Politi K, Gettinger SN, Wilson LD, Herbst RS, Patel AA. Early Assessment of Lung Cancer Immunotherapy Response via Circulating Tumor DNA. Clin Cancer Res. 2018 Apr 15;24(8):1872-1880. doi: 10.1158/1078-0432.CCR-17-1341. Epub 2018 Jan 12. PMID 29330207
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Background] Koch M, Garden OJ, Padbury R, Rahbari NN, Adam R, Capussotti L, Fan ST, Yokoyama Y, Crawford M, Makuuchi M, Christophi C, Banting S, Brooke-Smith M, Usatoff V, Nagino M, Maddern G, Hugh TJ, Vauthey JN, Greig P, Rees M, Nimura Y, Figueras J, DeMatteo RP, Buchler MW, Weitz J. Bile leakage after hepatobiliary and pancreatic surgery: a definition and grading of severity by the International Study Group of Liver Surgery. Surgery. 2011 May;149(5):680-8. doi: 10.1016/j.surg.2010.12.002. Epub 2011 Feb 12. PMID 21316725
- [Background] Rahbari NN, Garden OJ, Padbury R, Brooke-Smith M, Crawford M, Adam R, Koch M, Makuuchi M, Dematteo RP, Christophi C, Banting S, Usatoff V, Nagino M, Maddern G, Hugh TJ, Vauthey JN, Greig P, Rees M, Yokoyama Y, Fan ST, Nimura Y, Figueras J, Capussotti L, Buchler MW, Weitz J. Posthepatectomy liver failure: a definition and grading by the International Study Group of Liver Surgery (ISGLS). Surgery. 2011 May;149(5):713-24. doi: 10.1016/j.surg.2010.10.001. Epub 2011 Jan 14. PMID 21236455
- [Background] Leslie K, Troedel S, Irwin K, Pearce F, Ugoni A, Gillies R, Pemberton E, Dharmage S. Quality of recovery from anesthesia in neurosurgical patients. Anesthesiology. 2003 Nov;99(5):1158-65. doi: 10.1097/00000542-200311000-00024. PMID 14576554
- [Background] Myles PS, Weitkamp B, Jones K, Melick J, Hensen S. Validity and reliability of a postoperative quality of recovery score: the QoR-40. Br J Anaesth. 2000 Jan;84(1):11-5. doi: 10.1093/oxfordjournals.bja.a013366. PMID 10740540
- [Background] Shida D, Wakamatsu K, Tanaka Y, Yoshimura A, Kawaguchi M, Miyamoto S, Tagawa K. The postoperative patient-reported quality of recovery in colorectal cancer patients under enhanced recovery after surgery using QoR-40. BMC Cancer. 2015 Oct 26;15:799. doi: 10.1186/s12885-015-1799-3. PMID 26503497
- [Background] Peng LH, Wang WJ, Chen J, Jin JY, Min S, Qin PP. Implementation of the pre-operative rehabilitation recovery protocol and its effect on the quality of recovery after colorectal surgeries. Chin Med J (Engl). 2021 Nov 3;134(23):2865-2873. doi: 10.1097/CM9.0000000000001709. PMID 34732661
- [Background] Lee JH, Kim D, Seo D, Son JS, Kim DC. Validity and reliability of the Korean version of the Quality of Recovery-40 questionnaire. Korean J Anesthesiol. 2018 Dec;71(6):467-475. doi: 10.4097/kja.d.18.27188. Epub 2018 Apr 24. PMID 29684992
- [Background] Tanaka Y, Wakita T, Fukuhara S, Nishiwada M, Inoue S, Kawaguchi M, Furuya H. Validation of the Japanese version of the quality of recovery score QoR-40. J Anesth. 2011 Aug;25(4):509-15. doi: 10.1007/s00540-011-1151-2. Epub 2011 May 31. PMID 21626452
- [Background] McMillan DC, Crozier JE, Canna K, Angerson WJ, McArdle CS. Evaluation of an inflammation-based prognostic score (GPS) in patients undergoing resection for colon and rectal cancer. Int J Colorectal Dis. 2007 Aug;22(8):881-6. doi: 10.1007/s00384-006-0259-6. Epub 2007 Jan 24. PMID 17245566
- [Background] Shrotriya S, Walsh D, Bennani-Baiti N, Thomas S, Lorton C. C-Reactive Protein Is an Important Biomarker for Prognosis Tumor Recurrence and Treatment Response in Adult Solid Tumors: A Systematic Review. PLoS One. 2015 Dec 30;10(12):e0143080. doi: 10.1371/journal.pone.0143080. eCollection 2015. PMID 26717416
- [Background] Fruhling P, Hellberg K, Ejder P, Stromberg C, Urdzik J, Isaksson B. The prognostic value of C-reactive protein and albumin in patients undergoing resection of colorectal liver metastases. A retrospective cohort study. HPB (Oxford). 2021 Jun;23(6):970-978. doi: 10.1016/j.hpb.2020.10.019. Epub 2020 Nov 16. PMID 33214053
- [Background] Punt CJ, Buyse M, Kohne CH, Hohenberger P, Labianca R, Schmoll HJ, Pahlman L, Sobrero A, Douillard JY. Endpoints in adjuvant treatment trials: a systematic review of the literature in colon cancer and proposed definitions for future trials. J Natl Cancer Inst. 2007 Jul 4;99(13):998-1003. doi: 10.1093/jnci/djm024. Epub 2007 Jun 27. PMID 17596575
- [Background] Karanicolas PJ, Farrokhyar F, Bhandari M. Practical tips for surgical research: blinding: who, what, when, why, how? Can J Surg. 2010 Oct;53(5):345-8. No abstract available. PMID 20858381
- [Background] Tsai MS, Su YH, Ho MC, Liang JT, Chen TP, Lai HS, Lee PH. Clinicopathological features and prognosis in resectable synchronous and metachronous colorectal liver metastasis. Ann Surg Oncol. 2007 Feb;14(2):786-94. doi: 10.1245/s10434-006-9215-5. Epub 2006 Nov 14. PMID 17103254
- [Background] Lochan R, White SA, Manas DM. Liver resection for colorectal liver metastasis. Surg Oncol. 2007 Jul;16(1):33-45. doi: 10.1016/j.suronc.2007.04.010. Epub 2007 Jun 4. PMID 17544654
- [Background] Bismuth H, Chiche L. Surgery of hepatic tumors. Prog Liver Dis. 1993;11:269-85. No abstract available. PMID 8272515
- [Background] Soules MR, Sherman S, Parrott E, Rebar R, Santoro N, Utian W, Woods N. Executive summary: Stages of Reproductive Aging Workshop (STRAW). Climacteric. 2001 Dec;4(4):267-72. PMID 11770182
- See also: The Multiple Organ Dysfunction Syndrome. — http://www.ncbi.nlm.nih.gov/books/NBK6868/

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-08-19): https://cdn.clinicaltrials.gov/large-docs/13/NCT05677113/Prot_SAP_000.pdf